CLINICAL TRIAL: NCT01409980
Title: Triphalangeal Thumbs in the Pediatric Population: Long Term Outcomes Following Surgical Intervention
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Angela Wang, M.D., University of Utah
Other Study IDs: 49246
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Phalanx of Supernumerary Digit of Hand
Keywords: delta phalanx; thumb reconstructed; triphalangeal thumbs
MeSH Terms: conditions — Triphalangeal Thumb

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Triphalangeal Thumb: A search will be performed using CPT code 26587 (reconstruction of a supernumerary digit) at both Primary Children's Hospital and Shriners to identify all patients who Dr. Wang and Hutchinson operated on with a delta phalanx.

SUMMARY:
A triphalangeal thumb is a thumb with three phalanges. The thumb often appears long and fingerlike, and can sometimes be in the same plane as the other fingers. Anatomically, the extra phalanx can have different shapes. Several classification systems have been used, but the simplest and most often used is the Wood (1976) classification by the shape of the extra phalanx. If the extra phalanx is triangularly shaped it is classified as a type I. Type II has a rectangular shaped extra phalanx but it has not developed as a full phalanx. Type III is a full extra phalanx.

DETAILED DESCRIPTION:
A triphalangeal thumb is a thumb with three phalanges. The thumb often appears long and fingerlike, and can sometimes be in the same plane as the other fingers. Anatomically, the extra phalanx can have different shapes. Several classification systems have been used, but the simplest and most often used is the Wood (1976) classification by the shape of the extra phalanx. If the extra phalanx is triangularly shaped it is classified as a type I. Type II has a rectangular shaped extra phalanx but it has not developed as a full phalanx. Type III is a full extra phalanx.

Different treatment strategies have been developed based on the type of triphalangeal thumb. This project looks specifically at type I, or a delta phalanx. The goals of surgery in any type are to reconstruct the anatomic deformity with a stable, functional thumb while providing an acceptable appearance.

There is no consensus on how triphalangeal thumbs with a delta phalanx should be treated. Bunnell and Campbell in the 1940s advocated doing no surgery at all. Milch advocated excising the abnormal phalanx in the pediatric population but supporting non-operative treatment for the adult population. A potential unwanted result of excision has been an angulated joint. Buck-Gramcko proposed that excision of the delta phalanx combined with ligament reconstruction could give a better result than with excision alone.

Hovius recommended different treatment based on the age of presentation. For patients less than 6 years, he advocated excision of a transverse oval piece of skin, resection of the extra phalanx with reconstruction of the radial collateral ligament at the new IP joint, and lengthening of the ulnar collateral ligament. For patients older than 6 years, he advocates partial resection of the extra phalanx with correction of the angle and arthrodesis of the DIP joint. Usually, collateral ligament reconstruction is not necessary in these cases.

Horii et al reviewed 13 type I delta triphalangeal thumbs with no associated hand abnormalities. Surgical treatment for these patients consisted of excision of an accessory phalanx and the repair of the collateral ligament. The IP joint was temporarily fixed with Kirschner wires for 4-6 weeks. Mean follow-up was 8.9 years. All patients were satisfied with the improvement in appearance. The mean IP joint motion was 54 degrees. No patients complained of instability or pain in the IP joint. Only one patient had ten degrees of lateral bending. They recommend operating on these patients between ages 1-2 years, when the phalangeal epiphyses becomes clear. They felt that earlier excision allows for better joint adaptation. The children also will learn how to use their hands correctly.

Recently it has been debated that it is beneficial to wait to operate on these children until they are older, and their bones and joints have matured. At that point, an osteotomy could be performed. Although these results have not been published yet, several well-respected hand surgeons have concluded that their outcomes have been better on patients who have had delayed surgery.

In our institutions, children generally have their thumb reconstructed using a delta phalanx excision with repair of the ligament around 1 to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients under age 18 with a delta, or type I, phalanx
* Surgical intervention at Primary Children's Hospital or Shriners Hospital by Dr. Angela Wang or Dr. Douglas Hutchinson consisting of delta phalanx excision and ligament reconstruction

Exclusion Criteria:

* Patients with type II or III triphalangeal thumb
* Patients undergoing a secondary or revision surgery as their first surgery at our institutions

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A search will be performed using CPT code 26587 (reconstruction of a supernumerary digit) at both Primary Children's Hospital and Shriners to identify all patients who Dr. Wang and Hutchinson operated on with a delta phalanx.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
evaluate the long-term outcomes of surgical treatment for children treated at Primary Children's Medical Center and Shriners Hospital with a delta phalanx. | 1 year
  Outcomes being measured include objective measurements (stability of IP and MCP joints, ROM of IP and MCP joints, grip strength and key pinch) and subjective measurements (VAS for functionality, pain and appearance, and DASH).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Wang, M.D., Principal Investigator — University of Utah Orthopedic Center